CLINICAL TRIAL: NCT03901027
Title: The FAM-SOTC Intervention: Families of Children With Chronic Illnesses
Brief Title: FAM-SOTC Intervention for Families of Children With Chronic Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UIceland-12019EKS
Record Dates: First submitted 2019-03-20; First posted 2019-04-03 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Chronic Illnesses
Keywords: Parents; Children; Chronic Illnesses
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The effectiveness of the intervention was tested within a quasi-experimental study with one group pre- and-posttest design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents of children with chronic illnesses (Experimental): psycho-educational intervention for parents
  Interventions: Behavioral: Therapeutic Conversation Interventions

INTERVENTIONS:
Behavioral: Therapeutic Conversation Interventions — Parents (N=31) at the Children's Hospital at the National University Hospital of Iceland, got two sessions of the FAM-SOTC intervention focusing on emotional support, evidence based information and recommendations and on the strengths of family members. The parents meet with the Advanced Practice Nurse at the Children´s Hospital without the child in both sessions, but each session lasted for 45 to 90 minutes. The sessions were offered with 4-8 weeks interval.

SUMMARY:
Purpose: A growing number of families with children are dealing with chronic illnesses or health problems that places increased demand on the family. Nurses are in a core position to support and empower these families. The benefit of therapeutic conversation between nurses and families dealing with health problems have shown positive results and therefore received increasing attention. The aim of this study was to evaluate the benefits of two sessions of the Family Strength Oriented Therapeutic Conversation (FAM-SOTC) intervention, offered by advanced practice nurses (APN), for parents of children and adolescents with Juvenile idiopathic arthritis (JIA), epilepsy, diabetes, and with sleep disturbance with attention deficit hyperactivity disorder (ADHD).

Design: The effectiveness of the intervention was tested within a quasi-experimental study with one group pre- and-posttest design.

Method: The intervention was based on the Calgary family assessment and intervention models and the Illness Beliefs model and was offered in March 2015--December 2016. Parents (N=31) at the Children's Hospital at the National University Hospital of Iceland, got two sessions of the FAM-SOTC intervention focusing on emotional support, evidence based information and recommendations and on the strengths of family members.

DETAILED DESCRIPTION:
Sample Data were collected at the Children's Hospital (CH) at the National University Hospital of Iceland (NUHI) in Reykjavik, Iceland. The population of Iceland is about 340,000 people. The incidence of diabetes among children in Iceland is 18 per year, and similar frequency among children and adolescents is reported regarding arthritis, epilepsy and sleeping disorder with ADHD. Participants in this study were 31 primary caregivers who all were the mothers of the children/adolescents with diabetes, arthritis, epilepsy or sleeping disorder with ADHD (see Table 1). A research assistant offered all the primary caregivers (N = 39; n=38 mothers and n=1 father) of children with one of the above-mentioned illnesses/disorders at the time of the data collection, to participate in the study. The 31 primary caregivers, who signed the consent form, participated in the study and represented 80% response rate. Parents completed online the questionaires at the clinic, before they started the first session and then again after the second session. Three APN ,specialists in the child illness diagnosis and who had special graduate educational training in family system nursing or had a doctorate degree in family nursing, offered the families the FAM-SOTC intervention. The parents meet with the APN at the Children´s Hospital without the child in both sessions, but each session lasted for 45 to 90 minutes. The sessions were offered with 4-8 weeks interval.

Description of the FAM-SOTC intervention The description of the development of the FAM-SOTC as well as a figure of the FAM-SOTC intervention, has been published elsewhere.

The first FAM-SOTC session:

When the APN had greeted the parents and made them comfortable, a family assessment was conducted by drawing a family tree and the quality of the family relations indicated, as well as asking them who belonged to their family. Therapeutic questions were used and parents asked questions like where they got support from? The parents were encouraged to talk about their child's illness experience and to reflect on how they perceived the diagnose of the child/adolescent. Further, the main concerns of each of the parent where explored by using therapeutic questions such as: (a) What is your greatest challenge now? and (b) If something could be different, what would that be? Throughout the therapeutic conversaton's the nurse acknowledge the suffering of each family member and normalized their emotional responses. The nurse than drew attention to the family strengths that had been observed. Potential resources were then discussed and the nurse offered advice and education. At the end of the therapeutic conversations the nurse again mentioned the parents strengths and resources and a time was set for the next appointment.

The second FAM-SOTC session:

In the second session a revision was made from the first session. Parents were encouraged to talk about their experience and change in their daily life and how the chronic illness or disorder affected them and the family as a unit. In addition, therapeutic questions were used such as (a) What is the greatest challenge facing your family now? (b) Who in your family do you think the illness has the most impact on? (c) What has been most/less helpful for you to do, to cope with the illness diagnose(s)? The parents were told what the APN had learned from their conversation, from their strengths and from their concerns. Furthermore, the parents emotional responses were acknowledge by telling them that their feelings and worries were normal for parents of children with chronic illnesses/disorders who were in similar situations'. Potential resources for each family were identified. Information and advice was offered and before finishing this session, parents were reminded of taking care of their own health and well-being.

Procedures Data were collected from March 2015 to december 2016 using online LimeSurvey program (a professional online survey). The parents signed an informed consent which was provided by a clinical nurse specialist on each of the units, who participated in the study. The parents were given a code to login to online LimeSurvey where they could fill out the questionnaires.

Ethical approval Approval for the study was received from the Scientific Ethical Board of the participating hospital (39/2014). A notification of the study was sent to the National Bioethics Committee in Iceland (S7110).

ELIGIBILITY:
Inclusion Criteria:

* Being a parents of children/adolescents with diabetes, arthritis, epilepsy or sleeping disorder with ADHD who were in active treatment at a University Hospital.
* Parents needed to be fluent in the Icelandic language.

Exclusion Criteria:

* Parents who did not understand Icelandic or English.
* Parents who could not read or write at the 4th grade level.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The ICE-Perceived Family Support from nurses Questionnaire (14-Items) at baseline | 1 week
  Has two factors: Cognitive (alpha=0.874) and emotional (alpha=0.937) support. Total alpha= 0.952. Has been reported to be both reliable and valid. The range of the scores is between 1-5. The total scale score range from 14-70, with higher score indicating better outcome.
The ICE-Perceived Family Support from nurses Questionnaire (14-Items) | 8-10 weeks
  Has two factors: Cognitive (alpha=0.874) and emotional (alpha=0.937) support. Total alpha= 0.952. Has been reported to be both reliable and valid. The range of the scores is between 1-5. The total scale scores range from 14-70, with higher score indicating better outcome.
The ICE-Family Illness Beliefs Questionnaire (7-Items) at baseline | 1 week
  I a one factor instrument regarding families illness beliefs. Alpha=0.789-0.910. The instrument has been reported to be both reliable and valid. The range of the scores is between 1-5. The total scale score range from 7-35, with higher score indicating better outcome.
The ICE-Family Illness Beliefs Questionnaire (7-Items) | 8-10 weeks The total scale score range from 7-35, with higher score indicating better outcome.
  I a one factor instrument regarding families illness beliefs. Alpha=0.789-0.910. The instrument has been reported to be both reliable and valid. The range of the scores is between 1-5.

SECONDARY OUTCOMES:
the PedsQL-Family Impact Module (36-item) at baseline | 1 week
  The instrument assess the impact of pediatric chronic health conditions on parents and families. It includes 8 subscales regarding physical functioning, emotional functioning, social functioning, cognitive functioning, communications, worry, daily activities and family relationships. The instrument has been reported to be both valid and reliable and has been psychometrically tested with Cronbach's alpha of 0.970). The range of the scores is between 1-5. The total scale score range from 36-180, with higher score indicating better outcome.
the PedsQL-Family Impact Module (36-item) | 8-10 weeks
  The instrument assess the impact of pediatric chronic healht conditions on parents and families. It includes 8 subscales regarding physical functioning, emotional functioning, social functioning, cognitive functioning, communications, worry, daily activities and family relationships. The instrument has been reported to be both valid and reliable and has been psychometrically tested with Cronbach's alpha of 0.970). The range of the scores is between 1-5. The total scale score range from 36-180, with higher score indicating better outcome.
The PedsQL-Healthcare Satisfaction Generic Module (24-items) at baseline | 1 week
  The items are grouped into 6 domains associated with health care satisfaction: information, family inclusion, communication , technical skills, emotional needs and overall satisfaction. The instrument has been reported to be valid and has been psychometrically tested with cronbach´s alpha of 0.79. The range of the scores is between 1-5. The total scale score range from 24-120, with higher score indicating better outcome.
The PedsQL-Healthcare Satisfaction Generic Module (24-items) | 8-10 weeks
  The items are grouped into 6 domains associated with health care satisfaction: information, family inclusion, communication , technical skills, emotional needs and overall satisfaction. The instrument has been reported to be valid and has been psychometrically tested with cronbach´s alpha of 0.79. The range of the scores is between 1-5. The total scale score range from 24-120, with higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ása Þórisdóttir, Study Director — University of Iceland

IPD SHARING:
Plan to Share IPD: No